CLINICAL TRIAL: NCT04979039
Title: Heart Rate Variability Monitoring to Predict Hypotension Following Spinal Anesthesia for Cesarean Delivery: Prospective Observational Study
Brief Title: Heart Rate Variability to Predict Hypotension Following Spinal Anesthesia in Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Clinical professor, Seoul National University Bundang Hospital
Other Study IDs: HRV Csec Spinal HypoT
Record Dates: First submitted 2021-06-30; First posted 2021-07-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- normal pregnancy: Adult pregnant women scheduled for cesarean section under spinal anesthesia
  Interventions: Other: analgesia nociception index (ANI) monitoring

INTERVENTIONS:
Other: analgesia nociception index (ANI) monitoring — The ANI monitor starts lying on the bed in the waiting area before entering the operating room, and the monitoring period should be at least 15 minutes. After entering the operating room, monitoring begins again and is maintained during the operation.

SUMMARY:
Based on the patient's heart rate variability, the analgesia nociception index (ANI) measures the activity of the autonomic nervous system and the sympathetic/parasympathetic nervous system and expresses it as a numerical value through a specific algorithm. The investigators will analyze it and see if it has the ability to predict severe hypotension following spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult pregnant women scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Emergency cesarean section
* When performing general anesthesia or epidural anesthesia
* Multiple pregnancies
* Surgery in which massive hemorrhage and massive blood transfusion are expected due to placenta previa
* Cardiac arrhythmias, congestive heart failure, ischemic heart disease, congenital heart anomalies
* Cranial nervous system disease
* Autonomic nervous system-related underlying diseases not related to pregnancy
* Fetal malformations
* Those who have an allergic skin reaction to adhesive substances such as bandages

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult pregnant women scheduled for cesarean section under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
The change of averaged value | 15 min, 10 min and 5 min before entering the operating room; every 5 min after entering the operating room
  The change of averaged value presented in ANI monitor
The change of instantaneous value | 15 min, 10 min and 5 min before entering the operating room; every 5 min after entering the operating room
  The change of instantaneous value presented in ANI monitor
Total dose of injected phenylephrine | During the anesthesia (from initiation of anesthesia until the end of anesthesia)
Total dose of injected glycopyrrolate | During the anesthesia (from initiation of anesthesia until the end of anesthesia)
The change of systolic blood pressure | Every 1 min after entering the operating room until finishing the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea